CLINICAL TRIAL: NCT03180931
Title: Mechanisms of Very Late Bioresorbable Scaffold Thrombosis Assessed by Optical Coherence Tomography: Insights From the International INVEST Registry
Brief Title: Independent OCT Registry on Very Late Bioresorbable Scaffold Thrombosis
Acronym: INVEST
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: INVEST
Record Dates: First submitted 2017-05-31; First posted 2017-06-08 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Coronary Thrombosis; Tomography, Optical Coherence; Drug-Eluting Stents
MeSH Terms: conditions — Coronary Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Scaffold thrombosis: Any patients who suffered from scaffold thrombosis occurring beyond 1 year after implantation of a Absorb BVS 1.1 and investigated by OCT with sufficient image quality allowing for CoreLab analysis at the timepoint of thrombosis.
  Interventions: Device: Bioresorbable vascular scaffold

INTERVENTIONS:
Device: Bioresorbable vascular scaffold — No study specific procedures will be applied. Optical coherence tomography recordings at the time of very late scaffold thrombosis were obtained during clinical routine with one of the commercially available and approved optical coherence tomography consoles and catheters. The analysis will be conducted at the Core laboratory at Bern University Hospital, Bern, Switzerland using a systematic and validated approach.
  Every participant will be coded by getting a number (pseudonym) in the local institutes. In the Core Laboratory, data will be further coded to ensure anonymity of the participants.

SUMMARY:
Bioresorbable vascular scaffold (BVS, ABSORB BVS1.1, Abbott Vascular) has been approved (CE mark) and is used in daily clinical practice. While recent randomized controlled trials comparing BVS versus metallic drug-eluting stent showed higher risk of definite or probable device thrombosis after BVS implantation, the causes underlying thrombotic events occurring beyond one year after scaffold implantation remain unclear and require investigation in an independent manner.

The INVEST registry is a world-wide, multi-center, observational, retrospective, investigator-initiated registry, which will include any patients who suffered from very late (>1 year) scaffold thrombosis, underwent optical coherence tomography (OCT) at the time of thrombosis and provided informed consent for the further use of their health related data for this registry.

DETAILED DESCRIPTION:
Background: The 3-year clinical outcome data of ABSORB II study failed to reach the two co-primary endpoints of vasomotion and late loss, but also reported a higher risk of definite or probable stent thrombosis throughout 3 years (3% vs 0%, p=0.03) with the Absorb BVS compared with the metallic EES as well as myocardial infarction.(1) In addition, a numerically higher rate of definite very late device thrombosis (2% vs 0%, p=0.19) was observed. In ABSORB Japan study, malapposition and late strut discontinuities were observed at the timepoint of very late scaffold thrombosis in all the 4 cases of definite very late scaffold thrombosis.(2,3) There is mounting evidence from other studies with extended follow-up supporting the notion of an increased risk of very late scaffold thrombosis. While the causes of acute scaffold thrombosis are explained at least in part (i.e. underexpansion, increased strut thickness), the causes underlying thrombotic events occurring beyond one year after scaffold implantation remain unclear and require investigation in an independent manner.

The investigators have previously reported that scaffold discontinuity and restenosis during the resorption process may provide mechanistic explanations for very late scaffold thrombosis.(4) As this report was based on a limited number of cases, the investigators extend the OCT database to comprehensively study the phenomenon very late scaffold thrombosis.

Rationale: The investigators consider the establishment of an independent OCT registry of paramount important as more than 150 000 patients have been implanted with Absorb BVS worldwide. The findings may provide important insights to identify patients at increased risk in addition to considerations regarding long-term antiplatelet therapy.

Objectives: The specific aim is to systematically analyse scaffold thrombosis occurring beyond 1 year after implantation of a Absorb BVS 1.1 investigated by OCT at the timepoint of thrombosis (either prior or after thrombus aspiration).

Primary and secondary endpoint/outcome(s): The primary endpoint is the underlying main reason for stent thrombosis as per quantitative and qualitative analysis and per expert panel consensus. To investigate the underlying mechanisms of very late scaffold thrombosis, the investigators will systematically assess the following parameters:

* Distal and proximal reference area, mm2
* Scaffold area, mm2
* Lumen area, mm2
* Incomplete scaffold apposition area, mm2
* Neointimal area, mm2
* Intracoronary thrombus area, mm2
* Percent area stenosis, %
* Scaffold expansion, %
* Eccentricity index
* Presence of macrophage accumulations, %
* Uncovered struts, %
* Malapposed struts, %
* Neointimal thickness, µm
* Incomplete scaffold apposition distance, µm
* Thrombus area, mm2

Other study variables: Retrospective data about clinical and drugs history of patients, procedural features and any intracoronary imaging information will be collected and analysed. This will include data for any imaging information between index implantation and very late scaffold thrombosis, when available, in order to investigate the underlying mechanisms of very late scaffold thrombosis.

Inclusion Criteria:

1. Any patients who suffered from scaffold thrombosis occurring beyond 1 year after implantation of a Absorb BVS 1.1 and investigated by OCT at the timepoint of thrombosis.
2. Sufficient quality of the OCT recording allowing for CoreLab analysis.

Exclusion Criteria: No exclusion criteria will be applied.

OCT assessment: Commercially available ILUMIEN (St. Jude Medical) or OFDI (Terumo) system are used. The analysis will be conducted at the Core laboratory at Bern University Hospital, Bern, Switzerland using a systematic and validated approach.

The lumen contour is drawn by semi-automated detection using QCU-CMS software, following the endoluminal contour of the neointima with manual correction wherever required. In case of thrombus with low attenuation, the lumen contour can still be drawn. In case of high attenuation, the lumen contour was extrapolated when the lumen contour was visible in at least three quadrants. The scaffold area was measured by joining the middle points of the signal poor core of the abluminal side of the struts if at least one strut was clearly visible in every quadrant. Distal and proximal reference area and scaffold expansion were calculated as previously reported by the MUSIC (Multicenter Ultrasound Stenting in Coronaries) investigators.(5) The neointimal thickness is measured from the abluminal border of the black strut core to the lumen. Uncovered struts are defined in the absence of a homogenous coverage by neointima. If the apposed struts is not covered by neointima but rather by irregular tissue, struts are categorized as "apposed uncovered with superimposed thrombus". If the coverage of apposed struts cannot be assessed owing to the presence of attenuating thrombus precluding the evaluation of neointima, the struts were categorized as "apposed possibly uncovered". Malapposed struts were defined as struts where the abluminal surface was clearly separated from the vessel wall. Incomplete scaffold apposition (ISA) distance was measured from the abluminal border of the strut core to the vessel wall. If malapposed struts are partially or completely surrounded by thrombus, struts were regarded as malapposed with thrombus. The area between the backside of the struts and the vessel wall was measured as ISA area, while the neointimal area is measured as scaffold area - (lumen area - ISA area). Intracoronary thrombus was identified as any irregular mass inside the lumen, with a sharp border and various degrees of attenuation.

Angiography assessment: The analysis will be conducted at the Core laboratory at Bern University Hospital, Bern, Switzerland using a conventional quantitative coronary angiography software (Qangio XA).

Determination of sample size: Up a total number of 30 patients who suffered from very late scaffold thrombosis and underwent OCT will be analysed retrospectively. This sample size is justified by the need to have precise estimates of event rates in terms of narrow 95% confidence intervals.

Planned analysis: Descriptive statistics will be provided. The investigators will assess geographic association between distribution of thrombus within scaffold and abnormal findings assessed by OCT. Statistical analyses will be performed with R (R Foundation for Statistical Computing, Vienna, Austria). Continuous variables will be summarized as mean ± standard deviation or median ± 95% confidence interval, depending on normality of distribution. The investigators will assess underlying reasons for scaffold thrombosis based on the same methodology with previous publication.(6)

ELIGIBILITY:
Inclusion Criteria:

1. Any patients who suffered from scaffold thrombosis occurring beyond 1 year after implantation of a Absorb BVS 1.1 and investigated by OCT at the timepoint of thrombosis.
2. Sufficient quality of the OCT recording allowing for CoreLab analysis.

Exclusion Criteria:

* No exclusion criteria will be applied.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From the hospital records, any patients who fulfill the inclusion criteria will be retrospectively included in the study. To estimate the denominator, total number of patients who underwent Absorb BVS implantation will also be collected.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2016-12-02 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-07-25 (Actual)

PRIMARY OUTCOMES:
Underlying main reason for stent thrombosis | Baseline
  Underlying main reason for stent thrombosis per expert panel consensus

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz Räber, MD, PhD, Principal Investigator — Bern University Hospital; Stephan Windecker, MD, Principal Investigator — Bern University Hospital
Locations (19):
- 5th Medical Department with Cardiology, Kaiser Franz Josef Hospital, Vienna, Austria
- Department of Cardiology, University Hospital Leuven, Leuven, Belgium
- France (4):
  - Cardiology Department, CHU Clermont-Ferrand, Clermont-Ferrand
  - Department of Cardiology, University Hospital Caremeau, Nîmes
  - Department of Cardiology, CH F Mitterand, Pau Université Cedex, France., Pau
  - Department of Cardiovascular Medicine, Hypertension and Heart Failure Unit, Health Innovation Lab (Hi-Lab) Clinique Pasteur, Toulouse
- Germany (4):
  - Department of Cardiology, University of Giessen, Giessen
  - Department of Cardiology, Asklepios Klinik St. Georg, Hamburg
  - Heart Center, Segeberger Kliniken GmbH, Academic Teaching Hospital of the Universities of Kiel, Kiel
  - Deutsches Herzzentrum München, Technische Universität München,, Munich
- Hong Kong (2):
  - Cardiology Division, Department of Medicine, Pamela Youde Nethersole Eastern Hospital, Chai Wan
  - Cardiology Division, Department of Medicine, Queen Elizabeth Hospital, Kowloon
- Cardiology Division, Bolognini Hospital, Seriate, Italy
- Netherlands (3):
  - Academic Medical Center, University of Amsterdam, Amsterdam
  - Department of Cardiology, Thoraxcenter, Erasmus Medical Center, Rotterdam, the Netherlands., Rotterdam
  - Department of Cardiology, University Medical Centre Utrecht, Utrecht
- Cardiac Department, National University Heart Centre, Singapore, Singapore
- Hospital Universitari de Bellvitge, Institut d' Investigació Biomèdica de Bellvitge, Universitat de Barcelona, L' Hospitalet de Llobregat, Spain., Barcelona, Spain
- Department of Cardiology, Stadtspital Triemli, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Serruys PW, Chevalier B, Sotomi Y, Cequier A, Carrie D, Piek JJ, Van Boven AJ, Dominici M, Dudek D, McClean D, Helqvist S, Haude M, Reith S, de Sousa Almeida M, Campo G, Iniguez A, Sabate M, Windecker S, Onuma Y. Comparison of an everolimus-eluting bioresorbable scaffold with an everolimus-eluting metallic stent for the treatment of coronary artery stenosis (ABSORB II): a 3 year, randomised, controlled, single-blind, multicentre clinical trial. Lancet. 2016 Nov 19;388(10059):2479-2491. doi: 10.1016/S0140-6736(16)32050-5. Epub 2016 Oct 30. PMID 27806897
- [Background] Kimura T, Kozuma K, Tanabe K, Nakamura S, Yamane M, Muramatsu T, Saito S, Yajima J, Hagiwara N, Mitsudo K, Popma JJ, Serruys PW, Onuma Y, Ying S, Cao S, Staehr P, Cheong WF, Kusano H, Stone GW; ABSORB Japan Investigators. A randomized trial evaluating everolimus-eluting Absorb bioresorbable scaffolds vs. everolimus-eluting metallic stents in patients with coronary artery disease: ABSORB Japan. Eur Heart J. 2015 Dec 14;36(47):3332-42. doi: 10.1093/eurheartj/ehv435. Epub 2015 Sep 1. PMID 26330419
- [Background] Onuma Y, Sotomi Y, Shiomi H, Ozaki Y, Namiki A, Yasuda S, Ueno T, Ando K, Furuya J, Igarashi K, Kozuma K, Tanabe K, Kusano H, Rapoza R, Popma JJ, Stone GW, Simonton C, Serruys PW, Kimura T. Two-year clinical, angiographic, and serial optical coherence tomographic follow-up after implantation of an everolimus-eluting bioresorbable scaffold and an everolimus-eluting metallic stent: insights from the randomised ABSORB Japan trial. EuroIntervention. 2016 Oct 20;12(9):1090-1101. doi: 10.4244/EIJY16M09_01. PMID 27597270
- [Background] Raber L, Brugaletta S, Yamaji K, O'Sullivan CJ, Otsuki S, Koppara T, Taniwaki M, Onuma Y, Freixa X, Eberli FR, Serruys PW, Joner M, Sabate M, Windecker S. Very Late Scaffold Thrombosis: Intracoronary Imaging and Histopathological and Spectroscopic Findings. J Am Coll Cardiol. 2015 Oct 27;66(17):1901-14. doi: 10.1016/j.jacc.2015.08.853. PMID 26493663
- [Background] de Jaegere P, Mudra H, Figulla H, Almagor Y, Doucet S, Penn I, Colombo A, Hamm C, Bartorelli A, Rothman M, Nobuyoshi M, Yamaguchi T, Voudris V, DiMario C, Makovski S, Hausmann D, Rowe S, Rabinovich S, Sunamura M, van Es GA. Intravascular ultrasound-guided optimized stent deployment. Immediate and 6 months clinical and angiographic results from the Multicenter Ultrasound Stenting in Coronaries Study (MUSIC Study). Eur Heart J. 1998 Aug;19(8):1214-23. doi: 10.1053/euhj.1998.1012. PMID 9740343
- [Background] Taniwaki M, Radu MD, Zaugg S, Amabile N, Garcia-Garcia HM, Yamaji K, Jorgensen E, Kelbaek H, Pilgrim T, Caussin C, Zanchin T, Veugeois A, Abildgaard U, Juni P, Cook S, Koskinas KC, Windecker S, Raber L. Mechanisms of Very Late Drug-Eluting Stent Thrombosis Assessed by Optical Coherence Tomography. Circulation. 2016 Feb 16;133(7):650-60. doi: 10.1161/CIRCULATIONAHA.115.019071. Epub 2016 Jan 13. PMID 26762519
- [Derived] Yamaji K, Ueki Y, Souteyrand G, Daemen J, Wiebe J, Nef H, Adriaenssens T, Loh JP, Lattuca B, Wykrzykowska JJ, Gomez-Lara J, Timmers L, Motreff P, Hoppmann P, Abdel-Wahab M, Byrne RA, Meincke F, Boeder N, Honton B, O'Sullivan CJ, Ielasi A, Delarche N, Christ G, Lee JKT, Lee M, Amabile N, Karagiannis A, Windecker S, Raber L. Mechanisms of Very Late Bioresorbable Scaffold Thrombosis: The INVEST Registry. J Am Coll Cardiol. 2017 Nov 7;70(19):2330-2344. doi: 10.1016/j.jacc.2017.09.014. PMID 29096803